CLINICAL TRIAL: NCT02953301
Title: A Multicentre, Double Blind, Randomised, Placebo-controlled, Phase II Trial to Evaluate Resminostat for Maintenance Treatment of Patients With Advanced Stage (Stage IIB-IVB) Mycosis Fungoides (MF) or Sézary Syndrome (SS) That Have Achieved Disease Control With Systemic Therapy - the RESMAIN Study
Brief Title: Resminostat for Maintenance Treatment of Patients With Advanced Stage Mycosis Fungoides (MF) or Sézary Syndrome (SS)
Acronym: RESMAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 4SC AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4SC-201-6-2015; 2016-000807-99 (EudraCT Number)
Record Dates: First submitted 2016-10-26; First posted 2016-11-02 (Estimated); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous
Keywords: Cutaneous T-Cell Lymphoma (CTLC); Maintenance; resminostat; 4SC; HDAC; Mycosis Fungoides; Sézary Syndrome
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous | interventions — resminostat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- resminostat (Experimental): 3 x 200 mg tablets p.o., 5 days treatment followed by 9 days rest (cycles until progress or unacceptable toxicity)
  Interventions: Drug: resminostat
- Placebo (Placebo Comparator): 3 tablets p.o. matching verum, 5 days treatment followed by 9 days rest (cycles until progress or unacceptable toxicity)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: resminostat
  Other Names: 4SC-201
  Arms: resminostat
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether resminostat will be able to delay or prevent worsening of disease in patients with advanced stage mycosis fungoides or Sézary Syndrome that have recently achieved disease control with previous systemic therapy.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients with histologically confirmed MF (Stage IIB-IVB) or SS in an ongoing complete response (CR), partial response (PR) or stable disease (SD) after at least one prior systemic therapy according to local standards (including but not limited to α-interferon, bexarotene, total skin electron beam irradiation, chemotherapy) [the most recent systemic therapy must have been completed as planned or stopped due to unacceptable toxicity 2-12 weeks prior to randomisation]
* Eastern Cooperative Oncology Group (ECOG) status score 0-2
* Adequate haematological, hepatic and renal function

Main Exclusion Criteria:

* Patients with progressive disease (PD)
* Baseline corrected QT (QTc) interval > 500 milliseconds
* Concurrent use of any other specific anti-tumour therapy including psoralen photo chemotherapy (PUVA), chemotherapy, immunotherapy, hormonal therapy, radiation therapy, or experimental medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2024-08 (Actual)

PRIMARY OUTCOMES:
PFS (Progression-free survival) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, up to approximately 32 months
  The primary objective is to determine if maintenance treatment with resminostat increases progression free survival (PFS) compared to placebo in patients with advanced stage (Stage IIB-IVB) MF or SS that have achieved disease control (complete response [CR], partial response [PR] or stable disease [SD]) with previous systemic therapy.

SECONDARY OUTCOMES:
TTSW (Time to symptom worsening): pruritus | From date of randomisation to first date that criteria for symptom (pruritus) worsening have been met, up to approximately 32 months. Symptom worsening is defined as an increase of a minimum of 3 points on the visual analogue itching scale
  To determine if maintenance treatment with resminostat increases time to symptom (pruritus) worsening (TTSW) compared to placebo.

OTHER OUTCOMES:
TTP (Time to progression) | From date of randomization until the date of first documented progression, up to approximately 32 months
  Compare time to progression (TTP) in patients when treated with resminostat vs placebo
TTNT (Time to next treatment) | From date of randomisation to first date that new treatment is received, up to approximately 44 months.
  Compare time to next treatment (TTNT) in patients when treated with resminostat vs placebo
PFS2, PFS3 (Progression-free survival 2, 3) | From date of start of subsequent treatment to date of progression or death due to any cause in the absence of documented PD whilst receiving second and third line therapy, respectively, up to approximately 44 months
  Assess the effect of maintenance treatment with resminostat by means of PFS of subsequent treatments (PFS2, PFS3)
ORR (Overall response rate) | Percent of patients within each treatment Arm that achieve confirmed CR or PR relative to the number of patients belonging to the analysis population of interest, up to approximately 32 months.
  Compare overall response rate (ORR, including CR, PR) in patients when treated with resminostat vs placebo
DOR (Duration of response) | From date confirmed CR or PR (whichever is first) until the criteria for PD have been met, up to approximately 32 months.
  Compare duration of response (DOR) in patients when treated with resminostat vs placebo
OS (Overall survival) | From the day of randomisation to death from any cause, up to approximately 44 months.
  Compare overall survival (OS) in patients when treated with resminostat vs placebo
Incidence of treatment-related AEs and SAEs (Safety and tolerability) | Weekly for 3 cycles, then bi-weekly during treatment phase, up to approximately 9 months
  Assess the safety and tolerability of resminostat
HrQoL (Health related quality of life) | Every 28 days, up to approximately 32 months
  Compare changes in health related quality of life (HrQoL) parameters in patients when treated with resminostat vs placebo
Maximum Plasma Concentration [Cmax] | At Cycle 3, Day 1 at 0.75h, 2h and 4 h after intake of trial medication / at Cycle 3, Day 5 to be done pre-dose and at 2h and 7h after intake of trial medication
  Assess the maximum plasma concentration [Cmax] of resminostat and metabolites
Area Under the Curve [AUC] | At Cycle 3, Day 1 at 0.75h, 2h and 4 h after intake of trial medication / at Cycle 3, Day 5 to be done pre-dose and at 2h and 7h after intake of trial medication
  Assess the Area Under the Curve [AUC] of resminostat and metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Stadler, Prof., Principal Investigator — Johannes Wesling Klinikum, Minden, Germany
Locations (54):
- Austria (2):
  - Medizinische Universität Graz, Graz
  - Medizinische Universität Wien, Vienna
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitaire Ziekenhuizen, Leuven
- France (5):
  - Centre Hospitalier Universitaire (CHU) de Bordeaux - Hôpital Saint-André, Bordeaux
  - CHU Estaing, Clermont-Ferrand
  - Centre Hospitalier Lyon-Sud, Lyon
  - Chu Paris-Gh St-Louis Lariboisiere F.Widal Hopital, Paris
  - Hopital Robert Debre - CHU de Reims, Reims
- Germany (17):
  - Charité - Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum Bochum - St. Josef-Hospital, Bochum
  - Elbekliniken Buxtehude, Buxtehude
  - Uniklinik Köln, Cologne
  - Klinikum Dortmund, Dortmund
  - SRH Wald-Klinikum Gera, Gera
  - Universitätsmedizin Göttingen, Göttingen
  - Universitaetsklinikum Halle, Halle
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Schleswig-Holstein (UKSH), Campus Kiel, Kiel
  - HELIOS Klinikum, Krefeld
  - Klinikum der Stadt Ludwigshafen am Rhein, Ludwigshafen am Rhein
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsklinikum Mannheim, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - Universitäts-Hautklinik Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- ATTIKON Hospital and Cutaneous Lymphoma Clinic, Athens, Greece
- Italy (5):
  - Universita Di Firenze, Florence
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Universita Cattolica del Sacro Cuore, Roma
  - IFO San Gallicano, Rome
  - Ospedale Molinette, Turin
- Japan (5):
  - Niigata University Medical and Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Tohoku University Hospital, Sendai
  - Hamamatsu University School of Medicine, Shizuoka
  - University of Tsukuba Hospital, Tsukuba
- Leids Universitair Medisch Centrum (LUMC), Leiden, Netherlands
- Poland (4):
  - Medical University of Gdansk, Gdansk
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Uniwersytecki Szpital Kliniczny im. WAM - CSW, Lodz
  - Centrum Onkologii-Instytut im. Marii Sklodowskiej-Curie, Warsaw
- Spain (5):
  - Hospital Del Mar, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Uni. Nuestra Senora de Candelaria, Santa Cruz de Tenerife
  - Hospital General Universitario, Valencia
- Switzerland (3):
  - Centre hospitalier universitaire vaudois (CHUV), Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Universitätsspital Zürich, Zurich
- United Kingdom (4):
  - University Hospital, Birmingham
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St John's Institute Of Dermatology - Guy's & St Thomas' Nhs Foundation Trust, London
  - Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stadler R, Quaglino P, Woei-A-Jin FJSH, Dummer R, Mitteldorf C, Papadavid E, Ortiz Romero PL, Guenova E, Abe R, Cowan R, Bagot M, Dalle S, Fujimura T, Gambichler T, Morris S, Wehkamp U, Terheyden P, Cozzio A, Dippel E, Alberti-Violetti S, Romejko-Jarosinska J, Wozniacka A, Gonzalez Barca E, Pujol Vallverdu R, Ramelyte E, Bechter O, Suzuki K, Knobler R, Danhauser-Riedl S, Scarisbrick J; RESMAIN Investigators. Resminostat for maintenance treatment in patients with advanced-stage mycosis fungoides or Sezary syndrome: a multicentre, double-blind, randomised, placebo-controlled, phase 2 trial. Lancet Haematol. 2026 Feb;13(2):e98-e109. doi: 10.1016/S2352-3026(25)00322-9. PMID 41651641
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956